CLINICAL TRIAL: NCT03613259
Title: A Pilot Study Investigating ¹⁸F-FLT-PET as a Marker of Response to Preoperative Radiotherapy in Soft Tissue Sarcoma
Brief Title: Fluorothymidine F-18 PET in Diagnosing Patients With Intermediate or High Grade Soft Tissue Sarcoma
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Funding expired
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Arthur Hung, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00016373; NCI-2017-00833 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SOL-16169-LX; STUDY00016373 (Other: OHSU Knight Cancer Institute); P01CA042045 (NIH); P30CA069533 (NIH)
Record Dates: First submitted 2018-01-23; First posted 2018-08-03 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Stage II Adult Soft Tissue Sarcoma; Stage IIA Adult Soft Tissue Sarcoma; Stage IIB Adult Soft Tissue Sarcoma; Stage IIC Adult Soft Tissue Sarcoma; Stage III Adult Soft Tissue Sarcoma; Stage IV Adult Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — alovudine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (fluorothymidine F-18 PET) (Experimental): Patients receive fluorothymidine F-18 IV over 1 minute and undergo PET scan over 60 minutes 21 or less days prior to standard of care radiation therapy and 14 or less days prior to the standard of care surgery.
  Interventions: Drug: Fluorothymidine F-18; Other: Laboratory Biomarker Analysis; Procedure: Positron Emission Tomography

INTERVENTIONS:
Drug: Fluorothymidine F-18 — Given IV
  Other Names: ¹⁸F-FLT; 3'-deoxy-3'-(¹⁸F) fluorothymidine; 3'-deoxy-3'-[¹⁸F]fluorothymidine; fluorothymidine F 18
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Positron Emission Tomography — Undergo fluorothymidine F-18 PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; positron emission tomography scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This pilot early phase I trial studies how well fluorothymidine F-18 positron emission tomography (PET) works in imaging patients with intermediate or high grade soft tissue sarcoma. Fluorothymidine F-18 PET may provide useful information about the tumor's response to treatment and may give the doctors early results that would better help to plan the post-surgical therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine fluorothymidine F-18 (¹⁸F-FLT) uptake parameters before and after radiotherapy.

SECONDARY OBJECTIVES:

I. To correlate ¹⁸F-FLT uptake post-radiotherapy scan with pathologic response. II. To correlate levels the mitotic index in surgical specimens with the ¹⁸F-FLT uptake in post-radiation scans.

III. To correlate ¹⁸F-FLT uptake both pre- and post-radiotherapy with magnetic resonance imaging (MRI) enhancement both within and around the tumor.

TERTIARY OBJECTIVES:

I. To compare ¹⁸F-FLT uptake and fludeoxyglucose F-18 (FDG) uptake when FDG-PET-computed tomography (CT) is available, pre-radiation, post-radiation, or both.

II. To compare ¹⁸F-FLT uptake in post-radiation scans with local recurrences looking for spatial correlation.

OUTLINE:

Patients receive fluorothymidine F-18 intravenously (IV) over 1 minute and undergo PET scan over 60 minutes 21 or less days prior to standard of care radiation therapy and 14 or less days prior to the standard of care surgery.

After completion of study, patients are followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histological evidence of an intermediate or high grade soft tissue sarcoma (STS) of any stage
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension as >= 1 cm with CT scan or MRI
* Prior resection is allowed if there is measurable gross disease and the subject plans to have neoadjuvant radiotherapy followed by resection
* Eastern Cooperative Oncology Group (ECOG) performance status =< 4, Karnofsky performance status >= 40%
* Creatinine =< 3 x upper limit of normal (ULM)
* Blood urea nitrogen (BUN) =< 3 x ULN
* Participants should be willing and able to have both PET-CT scans
* Participants should be eligible for and plan to undergo neoadjuvant radiation therapy and should be seen by a radiation oncologist prior to beginning the study; radiation at an outside facility will be allowed
* Participants should be eligible for and plan to have resection with a surgeon specializing in STS at Oregon Health and Science University (OHSU) and should be seen by said surgeon prior to beginning the study
* Participants should have a life expectancy that is greater than the study duration
* Participants should be willing to use adequate contraception from the time of the first PET-CT scan to 2 months after radiotherapy finishes; should a woman become pregnant while participating in this study, she should inform her treating physician immediately
* Women with childbearing potential must have a negative pregnancy test before each PET-CT scan
* Participants should have the ability to understand and the willingness to sign a written informed consent document
* Participants must sign a study specific consent form prior to registration

Exclusion Criteria:

* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or significant inflammation at treatment site or psychiatric illness/social situations that would limit compliance with study requirements or whose lab values do not meet the criteria above are excluded
* Pregnant women are excluded from this study
* Breast feeding women are excluded from this study
* Patients receiving chemotherapy during the course of radiation are excluded
* Patients whose weights exceed the tolerance of the table are excluded; the weight limit at OHSU is 450 pounds (lbs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Fluorothymidine F-18 mean standardized uptake value (SUV) as response to therapy. | Pre (=< 21 days before radiation) and Post (=< 14 days before resection) radiation fluorothymidine F-18 positron emission tomography
  Measured by mean SUV where the response to therapy is Pathological Response Disease change in volume of tumor (in cm3) utilizing Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) with magnetic resonance imaging (MRI). Mean, median, standard deviation, and range will be reported for continuous variables. Box plot, histogram plot, and density plot may be used to graphically show the distribution of the continuous endpoints.

SECONDARY OUTCOMES:
Change in Fluorothymidine F-18 peak SUV as response to therapy | Pre (=< 21 days before radiation) and Post (=< 14 days before resection) radiation fluorothymidine F-18 positron emission tomography
  Measured by peak SUV value where the response to therapy is Pathological Response Disease change in volume of tumor (in cm3) utilizing Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) with magnetic resonance imaging (MRI). Mean, median, standard deviation, and range will be reported for continuous variables. Box plot, histogram plot, and density plot may be used to graphically show the distribution of the continuous endpoints.
Fluorothymidine F-18 mean SUV correlation with pathology mitotic index | Post (=< 14 days before resection) radiation fluorothymidine F-18 positron emission tomography
  Measured as Ki-67. Will assess the mitotic index of resection tissue. Spearman's correlation coefficient will be computed to assess the association between the mitotic index and fluorothymidine F-18 uptake parameters in post-radiation scans.
Fluorothymidine F-18 peak SUV correlation with pathology mitotic index | Post (=< 14 days before resection) radiation fluorothymidine F-18 positron emission tomography
  Measured as Ki-67. Will assess the mitotic index of resection tissue. Spearman's correlation coefficient will be computed to assess the association between the mitotic index and fluorothymidine F-18 uptake parameters in post-radiation scans.
Fluorothymidine F-18 peak SUV correlation with enhancement by MRI | Post (=< 14 days before resection) radiation fluorothymidine F-18 positron emission tomography
  Measured as Ki-67. Evaluated by the standard of care magnetic resonance imaging. Will assess the size and location of irregularly increased T2-weighted signal intensity. Descriptive statistical analysis will be conducted
Volume of T2 enhanced MRI | Pre (=< 21 days before radiation) and Post (=< 14 days before resection) radiation fluorothymidine F-18 positron emission tomography
  Measured in (cm3).

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Y Hung, MD, Principal Investigator — OHSU Knight Cancer Institute